CLINICAL TRIAL: NCT01320488
Title: Breast Cancer in Young Women: Is it Different?
Acronym: YoungWomen
Status: Suspended | Type: Observational
Why Stopped: Difficulty in enrolling patients
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC08/117
Record Dates: First submitted 2011-03-19; First posted 2011-03-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Female Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tumor and blood specimens to characterize the pathology and biology of the tumors, and establish tumor bank for future studies
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast cancer is the leading cancer among women in Saudi Arabia representing almost the third of cancer diagnosed in Saudi women. Breast cancer in Saudi women is more frequently observed at young age. The data on this observation is either lacking or scares. Furthermore, the pathological and molecular features of breast cancer in young women are not clear. The study will provide important information to the national health care planner about this disease in young women including shedding light on possible genetic risk factors

DETAILED DESCRIPTION:
The study is a prospective longitudinal cohort study of young women with breast cancer. Over a 3-year period, we aim to identify a total of 600 women with newly diagnosed breast cancer, of those 300 women age 40 and younger and 300 older women from academic and community health care institutions across the Riyadh area. It is anticipated at least 400 of these women will agree to participate in the study. The comparable control group of older patients with breast cancer will be used for study comparison. Patient surveys, medical record review, and blood and tissue collection will be utilized. Women will be surveyed every 6 months after diagnosis. The study will investigate short and long-term disease and treatment issues, and psychosocial concerns. We will also collect tumor and blood samples to characterize the pathological and molecular aspects of tumors, and establish tumor bank for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of breast cancer
* Age 40 or younger at diagnosis for study group and older women for control group
* Informed consent obtained from patient

Exclusion Criteria:

* Absence of informed consent

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed project is a prospective longitudinal cohort study of young women with breast cancer. Over a 3-year period, we aim to identify a total of 600 women with newly diagnosed breast cancer, of those 300 women age 40 and younger and 300 older women from academic and community health care institutions across the Riyadh area. It is anticipated that at least 400 of these women (from study and control group) will agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
experience of breast cancer in young women | 10 years
  To identify a cohort of young women (age 40 or younger) newly diagnosed with breast cancer in King Abdulaziz Medical City and other collaborating hospitals to assess a broad range of variables at baseline and over the course.

CONTACTS AND LOCATIONS:
Overall Officials: Omalkahir Abulkhair, MD, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia